CLINICAL TRIAL: NCT04890457
Title: Transcutaneous Vagus Nerve Stimulation Promotes Oxytocin Release and Increases Fixations on Nose
Brief Title: Brain, Behavior and Endocrine Effects of Transcutaneous Vagus Nerve Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-81
Record Dates: First submitted 2021-05-12; First posted 2021-05-18 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Healthy
Keywords: Transcutaneous vagus nerve stimulation; Oxytocin release; Eye-tracking

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tragus then earlobe stimulation (Experimental)
  Interventions: Device: Vagus nerve stimulation via tragus; Device: Sham stimulation via earlobe
- Earlobe then tragus stimulation (Experimental)
  Interventions: Device: Vagus nerve stimulation via tragus; Device: Sham stimulation via earlobe

INTERVENTIONS:
Device: Vagus nerve stimulation via tragus — The device will send stimulus intensity around 0.5mA via tragus in the left ear (based on participants' subjective report), delivered with a pulse width of 0.25 ms at 25 Hz. Stimulation will be active for 30 seconds, followed by a break of 30 seconds.
Device: Sham stimulation via earlobe — The device will send stimulus intensity around 0.5mA via earlobe in the left ear (based on participants' subjective report), delivered with a pulse width of 0.25 ms at 25 Hz. Stimulation will be active for 30 seconds, followed by a break of 30 seconds.

SUMMARY:
The main aim of the study is to investigate whether the transcutaneous vagus nerve stimulation(tVNS) promotes oxytocin release and the potential biomarkers of tVNS based on eye-tracking data

DETAILED DESCRIPTION:
A randomized, single-blinded, sham-controlled, within-subject, crossover design will be employed in this study. In a randomized order, a total of 54 healthy subjects will receive transcutaneous vagus nerve stimulation via tragus and sham stimulation vis earlobe in the left ear (interval between these two stimulations will be 1 week). Eye-tracking and behavioral data will be collected before and after 30 minutes of stimulation, saliva samples will be collected before and after 30 minutes of stimulation, and the end of the experiment.

Some personal traits will be assessed using different kinds of questionnaires, such as the Autism Spectrum Quotient(ASQ), Social Responsiveness Scale(SRS), State-Trait Anxiety Inventory (STAI), Beck's Depression Inventory(BDI), and Toronto Alexithymia Scale (TAS-20).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorders

Exclusion Criteria:

* history of head injury;
* pregnant, menstruating, taking oral contraceptives;
* medical or psychiatric illness.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Oxytocin release | After 30 min tragus stimulation
  Investigating the oxytocin release after vagus nerve stimulation via tragus based on saliva samples

SECONDARY OUTCOMES:
The relationship between oxytocin concentration and personal traits | through study completion, an average of half an year
  Analyzing the correlation between saliva oxytocin concentration and scores on different personal traits
Pupil size | After 30 min tragus stimulation
  Investigating whether vagus nerve stimulation via tragus will increase pupil diameter

CONTACTS AND LOCATIONS:
Overall Officials: Keith Kendrick, Dr., Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China, Chengdu, Sichuan, China